CLINICAL TRIAL: NCT05405465
Title: Effectiveness of Golimumab in Patients With Ulcerative Colitis: Results of a Real-life Study in Switzerland
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Golimumab Real-world study
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis; Flare Up, Symptom
Keywords: Golimumab; Ulcerative Colitis; TNF-inhibitors; Clinical Response; Clinical Remission
MeSH Terms: conditions — Colitis, Ulcerative; Symptom Flare Up

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UC patients with exposure to golimumab: The investigators retrospectively analyzed all ulcerative colitis patients from the Swiss IBD cohort study treated with golimumab.
  Interventions: Drug: Exposure to golimumab

INTERVENTIONS:
Drug: Exposure to golimumab — Retrospective chart review to assess patient related outcomes and objective measures of inflammation at baseline, 6-10 weeks, 6 months, 12 months.

SUMMARY:
TNF inhibitors have improved treatment options for patients with inflammatory bowel disease (IBD) and three TNF inhibitors, infliximab, adalimumab and golimumab are available for treatment of ulcerative colitis in Switzerland. However, these drugs have been tested under ideal conditions in randomized controlled trials. Real-world data are needed to complement this information. It is the aim of the investigators to study, whether patients with ulcerative colitis can be effectively treated with golimumab in a real world setting in Switzerland.

The investigators used data from the Swiss IBD cohort study (SIBDC) in Switzerland and identified all SIBDC patients with UC treated with Golimumab and performed a retrospective chart review. The investigators acquired patient reported outcomes and objective measures for inflammation at baseline, at 6-10 weeks and at 6 and 12 months after golimumab treatment. Primary endpoint was clinical response (i.e. meaningful improvement) at 6-10 weeks. Secondary endpoints were clinical response at 6 and 12 months and clinical remission (i.e. free of symptoms of disease).

DETAILED DESCRIPTION:
Ulcerative colitis patients from the Swiss IBD cohort study treated with golimumab were identified. The investigators performed a retrospective chart review and assessed patient reported outcomes and objective measures of inflammation to assess response and remission.

As clinical response in UC the investigators defined a composite end point of: Marked improvement in partial Mayo score AND improvement in one or more of the following parameters (acquired during chart review):

* Endoscopy data
* Ultrasonography
* Calprotectin (cut off 100microg/g)
* CRP
* Anemia resolution

Marked improvement was defined as: Clinical response based on partial Mayo Score (including physician global assessment): decrease in partial Mayo score ≥ 2 points and ≥ 30% from baseline and a decrease in rectal bleeding subscore ≥ 1 point or absolute rectal bleeding score ≤ 1. Improvement in lab work was defined as a reduction of the difference between baseline values and the next limit of normal by ≥ 30%. Improvement in endoscopy/ ultrasonography was defined as a reduction of colitis in the same technique compared to baseline substantiated by images (endoscopy) or measurements of diameter of the bowel wall.

As clinical remission in UC we defined normalization (i.e. absence of pathology) of patient reported outcomes (Frequency of stool, blood in stool) AND no evidence of residual disease activity in all of the following parameters:

* Endoscopy data
* Ultrasonography
* Calprotectin (cut off 100microg/g)
* CRP and anemia

ELIGIBILITY:
Inclusion Criteria:

* Patient of the Swiss IBD cohort study
* Diagnosis of ulcerative colitis
* Past treatment with golimumab (at least one dose)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the Swiss IBD cohort study with ulcerative colitis treated with golimumab.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Response at week 6-10 | 6-10 weeks after first golimumab dose
  Clinical response at week 6-10

SECONDARY OUTCOMES:
Response at 6 months | 6 months after first golimumab dose
  Clinical response at 6 months
Response at 12 months | 12 months after first golimumab dose
  Clinical response at 12 months
Remission at week 6-10 | 6-10 weeks after first golimumab dose
  Clinical remission at week 6-10
Remission at 6 months | 6 months after first golimumab dose
  Clinical remission at 6 months
Remission at 12 months | 12 months after first golimumab dose
  Clinical remission at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided